CLINICAL TRIAL: NCT02945904
Title: IS Metomidate PET-CT Superior to Adrenal Venous Sampling in Predicting Outcome From Adrenalectomy in Patients With Primary Hyperaldosteronism
Acronym: MATCH
Status: Completed | Type: Observational
Sponsor: Queen Mary University of London (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); WBIC), Cambridge. University of Cambridge Addenbrookes Hospital, Cambridge CB2 2QQ (Unknown); Robertson Centre for Biostatistics University of Glasgow Glasgow G12 8QQ (Unknown); Barts and the London School of Medicine and Dentistry W Smithfield London - City of London EC1A 7BE (Unknown)
Responsible Party: Sponsor
Other Study IDs: 011149
Record Dates: First submitted 2016-09-05; First posted 2016-10-26 (Estimated); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Primary Aldosteronism; Hyperaldosteronism
MeSH Terms: conditions — Hyperaldosteronism | interventions — Adrenalectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Following adrenalectomy tissue will be genotyped for somatic mutations in KCNJ5, ATP1A1, ATP2B3, CACNA1D, CTNNB1 and phenotyping by histological grading, gene expression and immunohistochemistry.
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: adrenalectomy — Unilateral adrenalectomy for Conn's adenoma

SUMMARY:
Purpose of this clinical trial is to improve prediction of outcomes from surgical intervention in patients with Primary aldosteronism, and evaluate the merits of non-invasive metomidate PET CT versus adrenal vein sampling in the diagnosis of surgically correctable aldosteronism.

DETAILED DESCRIPTION:
This is an observational multi-centre prospective cohort study which takes place within secondary and tertiary care. All participants will have the same two investigations performed in random order. These are as follows:

11C- metomidate PET CT This is a one-hour non-invasive study, prior to which participants are treated with dexamethasone for 3 days. A proportion of patients will have an additional 18F-CETO PET CT scan to measure concordance between the two PET CT scans.

Adrenal Vein Sampling This is an invasive investigation in which both adrenal veins are cannulated and blood collected for measurement of adrenal steroid hormones. Adrenocorticotrophic hormone (ACTH) is administered prior to AVS in order to ensure steroid hormone secretion during the procedure.

The investigators will standardise the start-time of treatment with spironolactone, which is first-choice treatment for participants with primary aldosteronism, in order that the pre-spironolactone blood pressure and biochemistry can be compared with subsequent measurements post-surgery, and the changes during the first month of spironolactone treatment can be used to assess their value in predicting response to surgery.

Sub-study of Repeat 11-C Metomidate PET CT before and after Spironolactone therapy

In order to determine whether it will be necessary for the start of spironolactone treatment to be delayed in all participants until after both investigations are completed, the investigators will perform a sub-study, early in MATCH, in which 6 patients have their PET CT repeated after at least 6 weeks treatment with spironolactone. (This is the conventional period of time for which spironolactone is withdrawn prior to AVS.)

Follow-up management and investigations The investigators anticipate ~50% of participants will be found on one or both investigations to have unilateral PA, and be recommended for adrenalectomy.

The primary outcome measurements will be at 6 months after surgery, or 9-12 months following MDT decision, in those who do not undergo surgery.

Primary outcomes:

The following primary outcomes will be analysed hierarchically, with each analysis being considered as part of the primary analysis if all preceding analyses demonstrate statistical significance at p<0.05. Otherwise, analyses of subsequent outcomes will be considered to be secondary analyses.

* Normalisation of ARR at 6 months, defined as

  * ARRactivity < 750 pmol/L per ng/ml/hr
  * ARRmass < 91 miU/L
* Change in BP (mean of at least 6 measurements from home monitoring, or mean of at least 2 measurements from clinic ) from baseline to 6 months.
* Cure of hypertension at 6 months. Definitions of biochemical and clinical success based on the PASO criteria (using on data available on eCRF) will be used.

Each primary outcome will be analysed in the subgroup of participants who undergo surgery. For each of the above outcomes, AVS and 11C-metomidate PET CT will be judged to be 'accurate' if it indicated unilateral disease and if normalisation of ARR, reduction in SBP or cure of hypertension (measured hierarchically, in turn) was achieved at 6 months post-surgery; or if it did not indicate unilateral disease and the above outcomes were not achieved.

Estimated differences in accuracy will be reported with 95% CI and p-value between 11C-metomidate PET CT and AVS. For cure of hypertension at 6 month, non-inferiority of 11C-metomidate PET CT will be declared if the lower limit of the above 95% CI is greater than -17%. Each measure of cure based on the PASO criteria (biochemical, clinical) will be analysed in turn. Superiority of 11-C metomidate PET CT will be declared if p<0.05 and the lower limit of the 95% CI is greater than 0%."

Secondary outcomes

The secondary outcomes are:

* Biochemical success (based on PASO criteria) at 6 months, analysed as a 3-level categorical variable (complete, partial, absent)
* Clinical success (based on PASO criteria) at 6 months, analysed as a 3-level categorical variable (complete, partial, absent)
* Change in serum Potassium from baseline to 6 months
* Change in ARRactivity or ARRmass from baseline to 6 months
* Change in home SBP and DBP from baseline to 6 months
* Change in clinic SBP and DBO from baseline to 6 months
* Change in blood levels of Troponin, Brain Natriuretic Peptide from baseline to 6 months
* Changes in cardiac MRI measures of heart structure, anatomy and blood flow from baseline to 6 months
* Change in quality of life measures from baseline to 6 months

Secondary (and Primary) outcomes will be compared between participants who underwent surgery and those who did not; for those who underwent surgery, between those for whom surgery was indicated by AVS only, 11C-metomidate PET CT only, or for both investigations.

The sample size calculation has been performed to permit detection of a significant influence on outcome where the smallest number of patients will be available. This is the group of patients in whom the two diagnostic techniques give discordant results, estimated to be ~20% of the total.

Recruitment of 140 patients across 3 centres over 3 years (<1/centre/month), assuming an estimated 10% dropout, and 50% proceeding to adrenalectomy, permits 90% power at alpha=0.01 of detecting superiority of metomidate vs AVS in predicting hierarchical primary outcomes. The 25 patient extension, on the same assumptions regarding dropouts and proportion proceeding to surgery, will also provide 90% power to show non inferiority of 11C-metomidate PET CT in relation to AVS, within a margin of 18%.

ELIGIBILITY:
Summary of eligibility criteria Inclusion Criteria

* Male or female: Age >18 yrs.
* Diagnosis of PHA based on current published Endocrine Society consensus guidelines (Funder et al 2016)

Patients will be enrolled/consented when they have had each of the following:

At least one paired measurement of plasma renin and aldosterone, measured off spironolactone/eplerenone, showing an elevated ARR. With

1. either a plasma aldosterone >190 pmol/L after saline infusion
2. or 'spontaneous hypokalemia + plasma renin below detection levels + plasma aldosterone > 550 pmol/L)' (as per Endocrine Society guidance, 2016)
3. or failure to suppress plasma aldosterone by 30% + persistent PRA suppression after oral administration of captopril (as per Endocrine Society guidance, 2016)

and a CT or MRI scan of the adrenals with probable or definite adenoma(s) within the last five years

Patients with elevated ARR can be put forward for consideration by the MDT as exceptional cases in whom spironolactone/eplerenone is not (fully) withdrawn, and/or saline suppression is not performed, IF:

1. Plasma Aldosterone > 450 pmol/L AND plasma renin <0.5 pmol/ml/hr (<9 mU/L) if measured on treatment with ACEI (Lisinopril >=20 mg or equivalent) or ARB (Losartan 100 mg or equivalent); OR
2. Age <40 AND definite adrenal adenoma on CT or MRI Patients whose CT/MRI does not show probable or definite adenoma must also be reviewed by MDT before enrolment/consent

Any exception to the above diagnostic criteria will be subject to approval by monthly MDT.

Exclusion Criteria

* Those patients who indicate that they are unlikely to proceed with surgery will not be recruited, because there will be no outcome change in blood pressure, restoration of normal renin/angiotensin physiology) against which to compare the accuracy of the two Investigations.
* Patients contraindicated for spironolactone or eplerenone therapy.
* Any patients continuing on beta-blockers or direct renin blockers .
* Patients with eGFR <30 ml/min/ or expected to have a reduction in eGFR<30ml/min on aldosterone antagonist therapy.
* Pregnant / breastfeeding females unable/unwilling to take secure contraceptive precautions whilst undergoing investigations.
* Patients unwilling/unable to take the dexamethasone required to prepare for a metomidate PET-CT scan.
* Patients unwilling to have both 11- C Metomidate PET CT scan and Adrenal Vein Sampling.
* Any illness, condition or drug regimen that is considered a contraindication by the PI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with primary aldosteronism
Sampling Method: Probability Sample
Enrollment: 190 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Normalisation of aldosterone renin ratio (ARR) | Baseline to 6 month Primary endpoint
  change in aldosterone- renin ratio for renin activity/renin mass
Mean home systolic blood pressure | Baseline to 6 month primary endpoint
  Changes in average home systolic blood pressures

SECONDARY OUTCOMES:
Biochemical success using PASO categorical criteria complete, partial or absent | Baseline to 6 month Primary endpoint
  correction of hypokalaemia and normalisation of aldosterone-to- renin ratio
Clinical success using PASO categorical criteria complete, partial or absent | Baseline to 6 month Primary endpoint
  Reduction in blood pressure and reduction anti-hypertensive medication
Normal range serum potassium levels | Baseline to 6 month Primary endpoint
  normalisation of low serum potassium
Change in Aldosterone - renin ratio renin activity/renin mass (ARR) | Baseline to 6 month Primary endpoint
  change of ARR
Change in home systolic and diastolic blood pressure | Baseline to 6 month Primary endpoint
  change in home blood pressure readings
Change in clinic systolic and diastolic blood pressures | Baseline to 6 month Primary endpoint
  change in clinic blood pressures
change in troponin, Brain naturetic pepetide | Baseline to 6 month Primary endpoint
  serum measurements for troponin , naturetic Peptide
change in cardiac MRI measurements | Baseline to 6 month Primary endpoint
  Cardiac MRI scan at baseline and primary endpoint visit.
Change in quality of life | Baseline to 6 month Primary endpoint
  change in quality of life measures.

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Mary University of London, City of London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Goodchild E, Wu X, Senanayake R, MacFarlane J, Argentesi G, Laycock K, Bashari WA, Cabrera CP, O'Toole SM, Salsbury J, Benu D, Lee YN, Chua ACN, Matson M, Koo B, Parvanta L, Hilliard N, Kosmoliaptsis V, Marker A, Berney DM, Drew K, Tan W, Foo R, Mein CA, Wozniak E, Kearney J, Savage E, Sahdev A, Bird N, Smith G, Hird M, Warnes V, Gillett D, Dawnay A, Adeyeye E, Aigbirhio F, McIntosh A, McConnachie A, Cruickshank JK, Cheow H, Gurnell M, Drake WM, Brown MJ. Molecular Imaging Versus Adrenal Vein Sampling for the Detection of Surgically Curable Primary Aldosteronism : A Prospective Within-Patient Trial. Ann Intern Med. 2025 Mar;178(3):336-347. doi: 10.7326/ANNALS-24-00761. Epub 2025 Mar 4. PMID 40030172
- [Derived] Wu X, Senanayake R, Goodchild E, Bashari WA, Salsbury J, Cabrera CP, Argentesi G, O'Toole SM, Matson M, Koo B, Parvanta L, Hilliard N, Kosmoliaptsis V, Marker A, Berney DM, Tan W, Foo R, Mein CA, Wozniak E, Savage E, Sahdev A, Bird N, Laycock K, Boros I, Hader S, Warnes V, Gillett D, Dawnay A, Adeyeye E, Prete A, Taylor AE, Arlt W, Bhuva AN, Aigbirhio F, Manisty C, McIntosh A, McConnachie A, Cruickshank JK, Cheow H, Gurnell M, Drake WM, Brown MJ. [11C]metomidate PET-CT versus adrenal vein sampling for diagnosing surgically curable primary aldosteronism: a prospective, within-patient trial. Nat Med. 2023 Jan;29(1):190-202. doi: 10.1038/s41591-022-02114-5. Epub 2023 Jan 16. PMID 36646800